CLINICAL TRIAL: NCT06731231
Title: SGLT2i in Diabetic Patients with Renal Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS 299/2024
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-03

CONDITIONS: Post-transplant Diabetes Mellitus
Keywords: transplantation; renal; DM; PTDM; SGLT2i
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Renal Transplantation patients who are DM pre-study / PTDM who don't take SGLT2i
- Intervention (Active Comparator): Renal Transplantation patients who are DM pre-study / PTDM who take SGLT2i
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are glucose lowering agents used in the treatment of type 2 DM by improving glycemic control, weight reduction, blood pressure control and albuminuria. the use of SGLT2i as a cardiorenal protective tool may be of particular value in renal transplant patients due to the risk of multiple comorbidities such as diabetes and hypertension. Recently, sodium-glucose transport protein 2 inhibitors (SGLT2i) emerged as a new class of therapeutics with beneficial effects on both cardiovascular (CV) and kidney outcomes in patients with diabetic kidney disease, nondiabetic proteinuric chronic kidney disease (CKD), and heart failure with and without diabetes in patients with native kidneys
  Arms: Intervention

SUMMARY:
Post-transplant diabetes mellitus (PTDM), previously known as New Onset Diabetes After Transplantation defined as the diagnosis of diabetes mellitus (DM) in a previously non-diagnosed diabetic person after transplantation. PTDM is a common and serious post-transplant complication that threatens graft survival, increases incidence of infection and development of cardiovascular complications

The primary objective of this study is to assess efficacy and safety of dapagliflozin in patients with post-transplantation diabetic patients

DETAILED DESCRIPTION:
Post-transplant diabetes mellitus (PTDM), previously known as New Onset Diabetes After Transplantation defined as the diagnosis of diabetes mellitus (DM) in a previously non-diagnosed diabetic person after transplantation. PTDM is a common and serious post-transplant complication that threatens graft survival, increases incidence of infection and development of cardiovascular complications (Pham et al., 2020). The reported incidence of PTDM in kidney transplant recipients is 4% to 25% with 2- to 4-fold increased risk of cardiovascular and infectious complications as mentioned, which lowers patient survival. (Ying et al., 2020)

Historically, PTDM has been variably defined as having random glucose level greater than 200 mg/dL, fasting glucose level greater than 140 mg/dL, or the need for insulin or oral hypoglycemic agents in the posttransplant period, although not widely used in clinical practice, oral glucose tolerance (OGTT) remains the gold standard for diagnosing PTDM. It should be noted that the algorithmic approach to the screening and diagnosis of PTDM is largely based on published kidney transplantation literature. However, it is speculated that the principles are relevant to all forms of solid organ transplantation (Sharif et al., 2000).

Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are glucose lowering agents used in the treatment of type 2 DM by improving glycemic control, weight reduction, blood pressure control and albuminuria. the use of SGLT2i as a cardiorenal protective tool may be of particular value in renal transplant patients due to the risk of multiple comorbidities such as diabetes and hypertension. Recently, sodium-glucose transport protein 2 inhibitors (SGLT2i) emerged as a new class of therapeutics with beneficial effects on both cardiovascular (CV) and kidney outcomes in patients with diabetic kidney disease, nondiabetic proteinuric chronic kidney disease (CKD), and heart failure with and without diabetes in patients with native kidneys

SGLT2i exert their protective effects through tubuloglomerular feedback and reduced intraglomerular pressure, glycosuria and altered metabolism, natriuresis and blood pressure control, and other additional diuretic and hematopoietic effects reduction which may provide unique benefits to improve cardiorenal outcomes in kidney transplant patients

Evidence concerning the efficacy and safety of SGLT2i post renal transplantation is limited. Many of the mechanisms by which SGLT2i exert their benefit stand to prove equally as efficacious or more so among kidney transplant recipients as they have in patients with CKD. However, safety concerns have excluded transplant recipients from all large randomized control trials, and clinicians and patients alike are left to wonder if the benefits of these amazing drugs outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

- Must be able to swallow tablets kidney transplant recipient post-transplant ≥3 months In patients with Type 2 DM HbA1c ≥6.5% (48 mmol/mol) Or Fasting plasma glucose ≥126 mg/dL (7.0 mmol/L) Ir 2-hour plasma glucose during 75-g OGTT ≥200 mg/dL (11.1 mmol/L) Random plasma glucose ≥200 mg/dL (11.1 mmol/L) estimated GFR ≥30 ml/min/1.73m^2 Able to provide written consent Clinical diagnosis of Alzheimer's Disease

Exclusion Criteria:

Insulin dependent diabetes Thyroid disease Presence of severe peripheral vascular disease (i.e., prior amputation, gangrene, non-healing ulcer or ischemic rest pain); Presence of any hyper-coagulable state or thrombosis in the 3 months prior to screening Presence of any vascular insult as stroke or transient ischemic attack in the 3 months prior to screening; Prior episode of graft pyelonephritis in the 1 month prior to screening; Episode of acute graft rejection in the 3 months prior to screening; Untreated urinary or genital tract infection; Severe hypoglycemia within 3 months of screening women who are lactating or pregnant Prior SGLT2i allergy or intolerance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control by SGLT2i in post renal transplantation diabetic patients | 6 months
  The primary outcome was the control of fasting blood sugar with no episodes of hypoglycemic attacks with reduction of HbA1c
Assessing SGLT2i-related side effects in the intervention arm in comparison to the control arm | 6 months
  serious adverse events and adverse events of interest that may lead to premature discontinuation,interruption, or dose reduction of the study drug. Adverse effects of interest include volume depletion, UTI and genital infections, acute rejection, major hypoglycemia,, potential diabetic ketoacidosis, adverse effects leading to amputations, or events increasing the risk of lower-limb amputations.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospital, Cairo, Egypt